CLINICAL TRIAL: NCT06841445
Title: A Multicenter, Randomized, Double-blind, Placebo- Parallel Controlled, Phase II Study to Evaluate the Efficacy and Safety of HRS9531 Tablet in Obese Subjects
Brief Title: Efficacy and Safety of HRS9531 Tablet in Obese Subjects
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS9531-T-201
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Chronic Management of Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A: HRS9531 Tablet (Experimental)
  Interventions: Drug: HRS9531 Tablet
- Treatment group B: HRS9531 Tablet (Experimental)
  Interventions: Drug: HRS9531 Tablet
- Treatment group C: HRS9531 Tablet (Experimental)
  Interventions: Drug: HRS9531 Tablet
- Treatment group D: HRS9531 Tablet Placebo (Placebo Comparator)
  Interventions: Drug: HRS9531 Tablet placebo

INTERVENTIONS:
Drug: HRS9531 Tablet — HRS9531 Tablet dose 1
  Arms: Treatment group A: HRS9531 Tablet
Drug: HRS9531 Tablet — HRS9531 Tablet dose 2
  Arms: Treatment group B: HRS9531 Tablet
Drug: HRS9531 Tablet — HRS9531 Tablet dose 3
  Arms: Treatment group C: HRS9531 Tablet
Drug: HRS9531 Tablet placebo — HRS9531 Tablet placebo
  Arms: Treatment group D: HRS9531 Tablet Placebo

SUMMARY:
To evaluate the efficacy of HRS9531 tablet compared with placebo in reducing body weight in obese subjects after 26 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent;
2. Male or female subjects, 18-65 years of age at the time of signing informed consent;
3. At screening visit, 28.0 ≤BMI≤ 40.0 kg/m2;
4. Diet and exercise control for at least 3 months before screening visit, and the weight change does not exceed 5% within the last 3 months;
5. Non-pregnant or lactating women. Fertile male and female (including partners) agree to use highly effective contraceptive methods.

Exclusion Criteria:

1. Uncontrollable hypertension;
2. Presence of - clinically significant lab or ECG results that may affect the evaluation of the efficacy or safety of the study drug at screening visit;
3. PHQ-9 score ≥15;
4. Medical history or illness that affects body weight;
5. History of diabetes;
6. Acute infection, acute trauma, or medium to large surgery within 1 month prior to screening;
7. History of severe cardiovascular and cerebrovascular diseases within 6 months prior to screening;
8. Any organ-system malignancies developed within 5 years;
9. Confirmed or suspected depression, bipolar disorder, suicidal tendencies, schizophrenia, or other serious mental illness;
10. History of alcohol and/or substance abuse or drug abuse;
11. Use of any medication or treatment that may have caused significant weight change within 3 months;
12. History of bariatric surgery;
13. Known or suspected hypersensitivity to trial product(s) or related products;
14. history of blood donation or blood loss in the 3 months before screening, or blood transfusion in the 2 months before screening;
15. Surgery is planned during the trial;
16. Mentally incapacitated or speech-impaired;
17. Acute or chronic hepatitis;
18. The investigators determined that other conditions were inappropriate for participation in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage Change from baseline in body weight after 26 weeks of treatment | after 26 weeks of treatment

SECONDARY OUTCOMES:
Proportion of subjects with weight loss of ≥5% from baseline in body weight after 26 weeks of treatment | after 26 weeks of treatment
Proportion of subjects with weight loss of ≥10% from baseline in body weight after 26 weeks of treatment | after 26 weeks of treatment
Proportion of subjects with weight loss of ≥15% from baseline in body weight after 26 weeks of treatment | after 26 weeks of treatment
Change from baseline in body weight after 26 weeks of treatment | after 26 weeks of treatment
Change from baseline in waist circumference after 26 weeks of treatment | after 26 weeks of treatment
Change from baseline in BMI after 26 weeks of treatment | after 26 weeks of treatment
Change from baseline in blood pressure after 26 weeks of treatment | after 26 weeks of treatment
Change from baseline in blood lipid after 26 weeks of treatment | after 26 weeks of treatment
Change from baseline in blood uric acid after 26 weeks of treatment | after 26 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided